CLINICAL TRIAL: NCT04431518
Title: The Steady-State Pharmacokinetics (PK) of Dolutegravir/Rilpivirine Fixed Dose Combination (FDC) in Patients With End Stage Renal Disease (ESRD) Requiring Hemodialysis (HD)
Brief Title: Pharmacokinetics of JULUCA in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Samir K. Gupta, MD, Professor of Medicine, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ViiV Healthcare IIS 1837
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: HIV/AIDS; ESRD
Keywords: HIV; ESRD; Hemodialysis; Pharmacokinetics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Kidney Failure, Chronic | interventions — dolutegravir, rilpivirine drug combination

STUDY DESIGN:
Intervention Model Description: Matched case-control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hemodialysis Group (Experimental): Receipt of JULUCA one pill per day up to 14 days
  Interventions: Drug: JULUCA 50Mg-25Mg Tablet
- Normal Renal Function Group (Active Comparator): Receipt of JULUCA one pill per day up to 14 days
  Interventions: Drug: JULUCA 50Mg-25Mg Tablet

INTERVENTIONS:
Drug: JULUCA 50Mg-25Mg Tablet — One dose of JULUCA will be taken daily for up to 14 days

SUMMARY:
This study will compare the pharmacokinetics of the component drugs in JULUCA, and HIV combination treatment pill, in HIV-negative patients who require hemodialysis with those with normal renal function.

DETAILED DESCRIPTION:
The pharmacokinetics (PK) of dolutegravir (DTG) and rilpivirine (RPV), the components of JULUCA, in patients with end stage renal disease (ESRD) requiring hemodialysis (HD) have not previously been adequately studied. It is possible that the PK of these drugs are affected by renal failure which may then compromise effectiveness and safety. This trial will rigorously assess the plasma PK and protein-binding of these two drugs in 10 HIV-negative patients requiring hemodialysis with 10 matched persons with normal renal function. All participants will receive JULUCA for up to 14 days and then undergo a 24 hour intensive PK evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Negative HIV antibody testing at screening.
2. For the ESRD requiring HD study group: ESRD requiring chronic hemodialysis for at least 6 months at an established center (not home dialysis).

   NOTE: The approximate date that hemodialysis was initiated should be reported, if known.

   For the normal renal function group: Estimated CrCl (using the Cockcroft-Gault equation) at screening ≥75mL/min.
3. Availability of alternative venous access (not used for dialysis) for the purpose of PK sampling.
4. The following laboratory values obtained within 30 days prior to study entry (obtained either at screening or done as part of routine clinical care):

   * AST (SGOT) and ALT (SGPT) less than or equal to ULN
   * Total bilirubin less than or equal to 1.5 x ULN
   * Hemoglobin greater than or equal to 8.0 mg/dL
5. A negative serum pregnancy test result at screening for all women of reproductive potential who have not reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation.
6. Males and females, age 18-65 years.
7. Ability and willingness of participant or legal guardian/representative to provide written informed consent.

Exclusion Criteria:

1. Known allergy or hypersensitivity to either dolutegravir or rilpivirine
2. Use of peritoneal dialysis.
3. Serious illnesses, other than ESRD, requiring systemic treatment and/or hospitalization within 30 days prior to the Screening Visit.
4. Known liver cirrhosis, unstable liver disease (presence of ascites, encephalopathy, coagulopathy, esophageal/gastric varices), Child-Pugh Class A, B, or C, or known biliary abnormalities (except for known Gilbert's syndrome or asymptomatic gallstones).
5. Hepatitis B surface antigen or hepatitis C antibody with detectable RNA at screening.
6. Known gastrointestinal disease that may lead to poor absorption of the study drugs.
7. Known hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
8. Any of the following gastrointestinal signs or symptoms of Grade ≥ 2 within 7 days prior to the Screening Visit or during study drug administration prior to the Intensive PK Study Visit:

   * nausea
   * vomiting
   * diarrhea
   * abdominal pain
9. Use of any of the following within 30 days of initiating study drug:

   * Medications known to appreciably inhibit or induce CYP3A enzymes, P-glycoprotein, or UGT1A1 or UGT1A4 enzymes (e.g., anticonvulsants such as carbamazepine, phenytoin, oxacarbamazepine; antimycobacterials such as rifampin, rifabutin and rifapentine; antifungal agents such as ketoconazole, fluconazole and itraconazole; verapamil, clarithromycin, erythromycin)
   * St. John's Wort, echinacea, grapefruits or grapefruit juice, garlic supplements, ginseng, golden seal, and milk thistle
   * Cancer chemotherapeutic agents
   * Investigational agents
   * Immunomodulators, including systemic steroids greater than or equal to 100 mg/day of prednisone (Note: Topical and inhaled corticosteroids are allowed.)
   * Dofetilide
   * Positive pre-study drug screen. Drugs that will be screened for include amphetamines, barbiturates, cocaine and phencyclidine (PCP). Active injected drug users will be excluded from this study.
10. Use of proton pump inhibitors within 7 days of initiating study drug (H2 blockers are permitted).
11. Pregnancy and/or breast-feeding.
12. Moderate to severe depression, defined as a PHQ-9 ≥ 10 at Screening.
13. Significant change (i.e., more than a 50% change) in tobacco smoking habit within 6 weeks prior to the Screening Visit. Participants who have recently stopped smoking should have stopped smoking more than 6 weeks prior to the Screening Visit. Participants who have recently started smoking should have started more than 6 weeks prior to the Screening Visit.
14. QTc interval greater than 500 msec at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Samir Gupta, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD will provided upon request and approval by the investigators or through online data repositories such as Figshare.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will become available after publication of the data, anticipated to be by July 2022.
Access Criteria: Fully available when posted to online repositories. Additional data upon request and approval by the study investigators. The financial sponsor will not have a role in this process.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemodialysis Group | Normal Renal Function Group | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [50 to 60] | 57.25 [53 to 60] | 57.375 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dolutegravir (DTG) Ctau
Description: Steady-state plasma Ctau for dolutegravir at the intensive study visit, which occurred between days 11 and 14
Time Frame: 0 to 24 hours post-dose on the intensive study visit
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Number analyzed (Participants) | 4 | 4
ng/mL | 1259 (447) | 1666 (415)

2. Primary Outcome: Rilpivirine (RPV) Ctau
Description: Steady-state plasma Ctau for rilpivirine at the intensive study visit, which occurred between days 11 and 14
Time Frame: 0 to 24 hours post-dose on the intensive study visit
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Number analyzed (Participants) | 4 | 4
ng/mL | 50 (17) | 77 (47)

3. Secondary Outcome: Safety of DTG
Description: The attributable grade 3 or 4 adverse events associated with use of DTG will be assessed during the study. Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. Grade 3 indicates a severe event, and Grade 4 indicates a potentially life-threatening event.
Time Frame: 30 days
Measure: Number; unit: Adverse Events
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Number analyzed (Participants) | 4 | 4
Adverse Events | 0 | 0

4. Secondary Outcome: DTG AUC
Description: Steady-state plasma AUC for dolutegravir at the intensive study visit, which occurred between days 11 and 14
Time Frame: 0 to 24 hours post-dose on the intensive study visit
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Number analyzed (Participants) | 4 | 4
h*ng/mL | 78095 (28979) | 75301 (23090)

5. Secondary Outcome: DTG Cmax
Description: Steady-state plasma Cmax for dolutegravir at the intensive study visit, which occurred between days 11 and 14
Time Frame: 0 to 24 hours post-dose on the intensive study visit
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Hemodialysis Group | Normal Renal Function Group
Number analyzed (Participants) | 4 | 4
ng/mL | 6346 (2593) | 5984 (2804)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Hemodialysis Group | Normal Renal Function Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemodialysis Group (N=4) | Normal Renal Function Group (N=4)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT04431518/Prot_SAP_003.pdf
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04431518/ICF_004.pdf